CLINICAL TRIAL: NCT06850168
Title: Clinical Investigation of a Novel Spectacle Lens on Slowing Down Juvenile Myopia Progression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WS10367
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Myopia
Keywords: Refractive error; Eye disease; Axial length; Myopia control
MeSH Terms: conditions — Myopia; Refractive Errors; Eye Diseases

STUDY DESIGN:
Intervention Model Description: This is a 2-year, randomized, double-masked, contralateral, exploratory clinical trial with the objective to evaluate the efficacy of two test lenses designed with passive red-light emission in the control of myopia progression. The subject starts by wearing standard SVL, designed with passive red-light emission in one eye, and standard SVL in the contralateral eye. After 1 year, the eye wearing SVL designed with passive red-light emission will be replaced with standard MCL, and the contralateral eye will be replaced with standard MCL designed with passive red-light emission. At the end of the 2-year period, each eye would be exposed to lenses designed with passive red-light emission for 1 year each. There will be a total of 11 study visits with follow-up periods at 6 months, 12 months, 18 months and 24 months.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): (Year 1) OD: SVL with passive red-light emission; OS: SVL (Year 2) OD: MCL; OS: MCL with passive red-light emission
  Interventions: Device: SVL; Device: SVL with passive red-light emission; Device: MCL; Device: MCL with passive red-light emission
- Group B (Experimental): (Year 1) OD: SVL; OS: SVL with passive red-light emission (Year 2) OD: MCL with passive red-light emission; OS: MCL
  Interventions: Device: SVL; Device: SVL with passive red-light emission; Device: MCL; Device: MCL with passive red-light emission

INTERVENTIONS:
Device: SVL — Dispensed to one eye in Year 1
Device: SVL with passive red-light emission — Dispensed to the contralateral eye in Year 1.
Device: MCL — Dispensed to one eye in Year 2 (if used SVL with passive red-light emission in Year 1).
Device: MCL with passive red-light emission — Dispensed to the contralateral eye in Year 2 (if used SVL in Year 1).

SUMMARY:
The goal of this exploratory clinical trial is to evaluate the efficacy and safety of a test spectacle lens (standard single vision lens (SVL) during first year, and standard myopia control lens (MCL) in second year), designed with passive red-light emission, for the control of myopia progression in myopic children age 6 to 11 years old, both male and female, with no systemic or ocular anomalies. The main question it aims to answer is:

Does the test spectacle lens designed with passive red-light emission provide significant myopia control effect to children?

Researchers will compare the standard SVL designed with passive red-light emission to SVL (first year) and MCL designed with passive red-light emission to MCL (second year) to see if the test spectacle lens work to slow down myopia progression.

Participants will:

* Wear the study spectacles
* Visit Essilor R&D Centre for follow-up sessions

ELIGIBILITY:
Inclusion Criteria:

* Children equal to or greater than 6 years old and less than 11 years at the time of signing informed consent.
* Corrected spherical equivalent refraction (SER) between -0.75 D and -5.00 D with astigmatism not more than 2.50 D.
* Difference in SER (Anisometropia) between two eyes should not exceed 1.00 D.
* Best corrected visual acuity better than or equal to +0.10 log MAR (20/25 or better with Snellen).
* Be in good general health, based on his/her and parent's/guardian's knowledge.
* Agree to wear spectacles for >12 hours/day and at least 6 days/week.
* Willingness and ability to participate in investigation for 2 years and attend scheduled visits.

Exclusion Criteria:

* Any ocular or systemic pathologies known to affect refractive status (e.g. keratoconus, diabetes, Down's syndrome etc.)
* Any binocular vision anomalies
* Amblyopia
* Use of prior myopia control treatment like specialized myopia control spectacles and contact lenses at least in the previous one month.
* Current use of ocular or systemic medications which, in the investigator's opinion, may significantly affect pupil size, accommodation or refractive state.
* Participation in any clinical investigation within 30 days of the baseline visit.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Axial Length | From baseline to 12 months
Change in Axial Length | From 12 months to 24 months

SECONDARY OUTCOMES:
Change in Spherical Equivalent Refraction | From baseline to 12 months
Change in Spherical Equivalent Refraction | From 12 months to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tan, Principal Investigator — Essilor R&D Centre Singapore
Locations (1):
- Essilor R&D Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang Y, Zhu Z, Tan X, Kong X, Zhong H, Zhang J, Xiong R, Yuan Y, Zeng J, Morgan IG, He M. Effect of Repeated Low-Level Red-Light Therapy for Myopia Control in Children: A Multicenter Randomized Controlled Trial. Ophthalmology. 2022 May;129(5):509-519. doi: 10.1016/j.ophtha.2021.11.023. Epub 2021 Dec 1. PMID 34863776
- [Background] Dong J, Zhu Z, Xu H, He M. Myopia Control Effect of Repeated Low-Level Red-Light Therapy in Chinese Children: A Randomized, Double-Blind, Controlled Clinical Trial. Ophthalmology. 2023 Feb;130(2):198-204. doi: 10.1016/j.ophtha.2022.08.024. Epub 2022 Aug 29. PMID 36049646